CLINICAL TRIAL: NCT03517683
Title: A Randomized Clinical Trial for the Influence of Injection Rate of Intrathecal Mixture of Local Anesthesia on Hypotension in Cesarean Section
Brief Title: Influence of Injection Rate of Intrathecal Mixture of Local Anesthesia on Hypotension in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24032016
Record Dates: First submitted 2018-04-19; First posted 2018-05-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low speed (Experimental): Patients will receive intrathecal injection of the anesthetic mixture in a slow speed (1ml in 15 seconds)
  Interventions: Other: Low speed
- High speed (Active Comparator): Patients will receive intrathecal injection of the anesthetic mixture in a high speed (1ml in 5 seconds)
  Interventions: Other: High speed

INTERVENTIONS:
Other: Low speed — Speed of intrathecal injection will be 1ml in 15 seconds
  Arms: Low speed
Other: High speed — speed of intrathecal injection will be 1ml in 5 seconds
  Arms: High speed

SUMMARY:
Hypotension is the most common complication of neuraxial anesthesia in obstetric patients and its prevalence in cesarean section is about 50-90%. Maternal hypotension causes unpleasant symptoms such as nausea, vomiting, loss of consciousness, respiratory depression, and cardiac arrest. Hypotension may reduce placental perfusion and result in fetal acidosis and neurological injury. Several techniques have been proposed to prevent hypotension.

The recommended spinal block height to ensure patient comfort for Cesarean delivery is T4-6. Clinically, it is desirable that the spread of local anesthetic through the cerebrospinal fluid (CSF) achieves a sensory level no higher than the T4 dermatome to avoid extensive sympathetic block. It is also important that the spinal block level be no lower than T6 to avoid patient discomfort during peritoneal manipulation and uterine exteriorization. The effect of injection speed on spread of spinal anesthesia is controversial. Several studies have demonstrated more extensive spread with faster injection while others report either greater spread with slower injection, or no difference. Slow injection of hyperbaric bupivacaine 10 mg over 60 and 120 sec has been shown to reduce the incidence and severity of hypotension during Cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
Patients admitted to undergo elective c-section under spinal anesthesia will be randomized using the sealed envelope technique to Group I who will receive intrathecal injection in a slow speed 1ml in 15 sec and group II who will receive 1ml in 5 sec.

The baseline pulse rate, blood pressure, respiratory rate, and oxygen saturation will be recorded intraoperatively. The presence of preoperative hypotension, nausea and vomiting, and level of block at 5 and 10 mins post intrathecal injection will be assessed .

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiology physical status 1 and 2
* and scheduled for elective c-section surgery under spinal anesthesia

Exclusion Criteria:

* Patients with cardiac and psychological problems
* Patients who take sedatives or narcotics

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | within one hour
  demonstrate the effect of the injection speed (high and low) of the anesthesia mixture intrathecally on the incidence of hypotension measured through mean arterial pressure

SECONDARY OUTCOMES:
block level | 5 and 10 minutes after performing the injection
  demonstrate the effect of the injection speed on the level of block at 5 and 10 minutes
Number of participants experiencing nausea and vomiting | within one hour
  demonstrate the effect of the injection speed on nausea/vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon